CLINICAL TRIAL: NCT02482428
Title: A Randomized, Vehicle Controlled, Active Comparator, Parallel Group Study to Evaluate Efficacy, Safety, and Tolerability of Topical LFX453 Formulations in Patients With External Genital Warts (EGWs)
Brief Title: Efficacy and Tolerability of Topical LFX453 for External Genital Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLFX453X2202
Record Dates: First submitted 2015-05-26; First posted 2015-06-26 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: External Genital Warts
Keywords: human papilloma virus (HPV), Genital Warts, Sexually transmitted disease (STD), viral disease
MeSH Terms: conditions — Papillomavirus Infections; Condylomata Acuminata; Sexually Transmitted Diseases; Virus Diseases | interventions — Therapies, Investigational; Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LFX453 0.1% NMC (Experimental): LFX453 0.1% nanomedicinal cream (NMC) Twice daily applications for a maximum of 12 weeks
  Interventions: Drug: Investigational Treatment
- LLFX453 0.15% LCC (Experimental): LFX453 0.15% liquid crystal cream (LCC) Twice daily applications for a maximum of 12 weeks
  Interventions: Drug: Investigational Treatment
- Vehicle to NMC (Placebo Comparator): Vehicle to nanomedicinal cream (NMC) Twice daily applications for a maximum of 12 weeks
  Interventions: Drug: Investigational Treatment
- Vehicle to LCC (Placebo Comparator): Vehicle to liquid crystal cream (LCC) Twice daily applications for a maximum of 12 weeks
  Interventions: Drug: Investigational Treatment
- Aldara (Active Comparator): Aldara 5% cream 3 applications per week for a maximum of 16 weeks
  Interventions: Drug: Aldara

INTERVENTIONS:
Drug: Investigational Treatment — Applied twice daily for up to 12 weeks
  Arms: LFX453 0.1% NMC; LLFX453 0.15% LCC; Vehicle to LCC; Vehicle to NMC
Drug: Aldara — Applied 3 times a week for 16 weeks
  Other Names: imiquimod
  Arms: Aldara

SUMMARY:
The LFX453X2202 study tested the investigational drug LFX453 against placebo for safety, tolerability, and efficacy in treating genital warts in circumcised men, in parallel with an additional open label arm using imiquimod 5%.

During the study the patients received either LFX453, placebo or active comparator and the tolerability and safety was assessed continuously through local tolerability assessments and adverse event recorded. Efficacy was clinical evaluations and lesion count. During the study biopsies were taken for analysis of pharmacokinetics and biomarkers. Blood samples were taken for safety, pharmacokinetics (PK), and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Circumcised male 18-60 years
* Clinical diagnosis of external genital warts
* Agree to remain abstinent or to use condoms during intercourse for the duration of the study
* Agree to digital photographs of treated area

Exclusion Criteria:

* Any treatment of genital warts within one month of treatment start
* HPV vaccination
* presence of warts larger than 200 mm2
* Genital herpes within one month of treatment start
* History of Bowenoid papulosis
* significant illness within 2 weeks of treatment start
* use of other investigational drugs
* known hypersensitivity to study drugs or constituents
* history of ECG abnormalities
* History of significant heart conditions
* Impaired renal function
* Abnormal liver function
* History of immunodeficiency disease
* Drug or alcohol abuse
* Immunosuppressive therapies
* Malignancies in the past 5 years
* hypertrophic scarring

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 88 patients were randomized and treated in the study
Groups:
- LFX453 0.15% LCC: LFX453 0.15% liquid crystal cream (LCC) Twice daily applications for a maximum of 12 weeks
Period: Overall Study
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara
Started | 24 | 22 | 10 | 10 | 22
Completed | 15 | 10 | 9 | 8 | 15
Not Completed | 9 | 12 | 1 | 2 | 7
Not completed — Lost to Follow-up | 4 | 9 | 1 | 2 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — protocol deviation | 1 | 1 | 0 | 0 | 0
Not completed — subject/guardian decision | 4 | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara | Total
Number analyzed (Participants) | 24 | 22 | 10 | 10 | 22 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (10.15) | 33.3 (9.31) | 35.2 (6.75) | 38.1 (9.62) | 36.0 (9.59) | 35.3 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 24 | 22 | 10 | 10 | 22 | 88

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance of Disease at Week 14
Description: Number of participants achieving complete clearance of genital warts at Week 14
Time Frame: Week 14
Population: Pharmacodynamics (PD) data sets included all randomized patients For efficacy end points only there were combined analysis of the 2 vehicle groups. Vehicle groups were analyzed separately for safety and tolerability only.
Measure: Number; unit: participants
Groups:
- Combined Vehicle: Vehicle to nanomedicinal cream (NMC) and Vehicle to liquid crystal cream (LCC) Twice daily applications
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 15 | 10 | 17 | 16
participants | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: LFX453 0.1% NMC vs Combined Vehicle; Test type: Non-Inferiority or Equivalence — p value is provided; p = 0.862, Posterior mean; Mean Difference (Net) = 0.05, 90% CI 2-sided [-0.03 to 0.20], Standard Deviation 0.07
Statistical Analysis 2: Comparison: LFX453 0.15% LCC vs Combined Vehicle; Test type: Non-Inferiority or Equivalence — p value is provided; p = 0.541, posterior mean; Mean Difference (Net) = 0.02, 90% CI 2-sided [-0.07 to 0.19], Standard Deviation 0.07

2. Primary Outcome: Number of Adverse Events (AE)/Serious Adverse Events (SAE) as a Measure of Safety and Tolerability up to 30 Weeks
Description: Number of participants with at least one AE/SAE in the category up to 30 weeks
Time Frame: 30 weeks
Population: The safety analysis set included all patients that received any study drug. For Safety & Tolerability only the 2 vehicles have separate analysis.
Measure: Number; unit: participants
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara
Number analyzed (Participants) | 24 | 22 | 10 | 10 | 22
participants
  Adverse Events (AEs) | 3 | 5 | 3 | 2 | 10
  Serious Adverse Events (SAEs) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants That Had Partial Clearance Rate of at Least 75 Percent Reduction in External Genital Wart (EGW)s Count at End of Treatment (EOT) Week 12 or 16
Description: Number of Participants that had partial clearance rate of at least 75 percent reduction in External Genital Wart (EGW)s count at end of treatment (EOT) Week 12 or 16
Time Frame: End of Treatment (EOT) Week 12 or Week 16
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 16 | 10 | 17 | 14
participants | 2 | 1 | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/10 | 0/10 | 0/22
Other Adverse Events (participants affected / at risk) | 3/24 | 5/22 | 3/10 | 2/10 | 10/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LFX453 0.1% NMC (N=24) | LFX453 0.15% LCC (N=22) | Vehicle to NMC (N=10) | Vehicle to LCC (N=10) | Aldara (N=22)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
COELIAC DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
APPLICATION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 0 | 2
APPLICATION SITE PAIN (General disorders) | 0 | 0 | 0 | 0 | 1
APPLICATION SITE PRURITUS (General disorders) | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
TINEA CRURIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
AMYLASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1
CARDIAC MURMUR (Investigations) | 0 | 1 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
HAEMOGLOBIN URINE (Investigations) | 0 | 0 | 0 | 1 | 0
LIPASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
SLEEP DISORDER DUE TO GENERAL MEDICAL CONDITION, INSOMNIA TYPE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
GLYCOSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
GENITAL RASH (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
PRURITUS GENITAL (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
SCROTAL ERYTHEMA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
SCROTAL ULCER (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.